CLINICAL TRIAL: NCT04500171
Title: Colorectal Cancer Screening Assessment Study in American Samoa
Brief Title: Colorectal Cancer Screening Assessment Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Cassel-2020-1
Record Dates: First submitted 2020-07-23; First posted 2020-08-05 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer
Keywords: health literacy; screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The health belief model and social cognitive theory were used as foundational principles to develop an intervention that builds awareness to initiate a CRC screening behavior modification.
  This research project will be the first to test the efficacy of the ColoCare FOBT home kit as a CRC screening intervention using a classical experimental (randomized clinical trial) in American Samoa. Second, the ColoCare kits can be identified as a cost-effective and culturally appropriate alternative to traditional FOBT home test kits. Lastly, results will be used to develop recommendations in healthcare delivery systems to improve information, communication, informed decision-making, and access to care in American Samoa.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- English Original Assessment Tools (Active Comparator): Short-Test of Functional Health Literacy in Adults ColoCARE Instruction Sheet CDC Colorectal Cancer Screening for Life Brochure ColoCARE Reply Card
  Interventions: Behavioral: Colocare Instruction Sheet: SAM + CAM SMOG; Behavioral: CDC Colorectal cancer screening for life brochure: SAM + CAM SMOG
- Samoan Original Assessment Tools (Active Comparator): Samoan Short-Test of Functional Health Literacy in Adults ColoCARE Instruction sheet CDC Colorectal Cancer Screening for Life Brochure ColoCARE Reply Card
  Interventions: Behavioral: Colocare Instruction Sheet: SAM + CAM Cloze Procedure; Behavioral: CDC Colorectal cancer screening for life brochure: SAM + CAM Cloze Procedure
- English Modified Assessment Tools (Experimental): Short-Test of Functional Health Literacy in Adults Modified ColoCARE Instruction Sheet Modified Colorectal Cancer Screening Brochure ColoCARE Reply Card
  Interventions: Behavioral: Colocare Instruction Sheet: SAM + CAM - Superior rating SMOG - 5th Grade Level; Behavioral: CDC Colorectal Cancer Screening for Life Brochure: SAM + CAM - Superior rating SMOG - 5th Grade Level; Behavioral: Colocare Instruction Video: Modified SAM + CAM -Superior rating
- Samoan Modified Assessment Tools (Experimental): Samoan Short Test of Functional Health Literacy in Adults Modified ColoCARE Instruction Sheet Modified Colorectal Cancer Screening Brochure ColoCARE Reply Card
  Interventions: Behavioral: Colocare Instruction Video: Modified SAM + CAM -Superior rating; Behavioral: Colocare Instruction Sheet: SAM + CAM - Superior rating Cloze Procedure; Behavioral: CDC Colorectal Cancer Screening for Life Brochure: SAM + CAM - Superior rating Cloze Procedure

INTERVENTIONS:
Behavioral: Colocare Instruction Sheet: SAM + CAM SMOG — Suitability and Comprehensibility Assessment of Materials (SAM + CAM). The SAM + CAM is comprised of 22 evaluation items within the 6 original categories. The SMOG is a readability assessment tool that uses a formula to calculate grade levels by the number of sentences, total number of words in the sentences, and the number of polysyllabic words
  Arms: English Original Assessment Tools
Behavioral: CDC Colorectal cancer screening for life brochure: SAM + CAM SMOG — Suitability and Comprehensibility Assessment of Materials (SAM + CAM). The SAM + CAM is comprised of 22 evaluation items within the 6 original categories. The SMOG is a readability assessment tool that uses a formula to calculate grade levels by the number of sentences, total number of words in the sentences, and the number of polysyllabic words
  Arms: English Original Assessment Tools
Behavioral: Colocare Instruction Sheet: SAM + CAM - Superior rating SMOG - 5th Grade Level — Suitability and Comprehensibility Assessment of Materials (SAM + CAM). The SAM + CAM is comprised of 22 evaluation items within the 6 original categories. The SMOG is a readability assessment tool that uses a formula to calculate grade levels by the number of sentences, total number of words in the sentences, and the number of polysyllabic words
  Arms: English Modified Assessment Tools
Behavioral: CDC Colorectal Cancer Screening for Life Brochure: SAM + CAM - Superior rating SMOG - 5th Grade Level — Suitability and Comprehensibility Assessment of Materials (SAM + CAM). The SAM + CAM is comprised of 22 evaluation items within the 6 original categories. The SMOG is a readability assessment tool that uses a formula to calculate grade levels by the number of sentences, total number of words in the sentences, and the number of polysyllabic words
  Arms: English Modified Assessment Tools
Behavioral: Colocare Instruction Video: Modified SAM + CAM -Superior rating — Suitability and Comprehensibility Assessment of Materials (SAM + CAM). The SAM + CAM is comprised of 22 evaluation items within the 6 original categories. The SMOG is a readability assessment tool that uses a formula to calculate grade levels by the number of sentences, total number of words in the sentences, and the number of polysyllabic words
  Arms: English Modified Assessment Tools; Samoan Modified Assessment Tools
Behavioral: Colocare Instruction Sheet: SAM + CAM Cloze Procedure — Suitability and Comprehensibility Assessment of Materials (SAM + CAM). The SAM + CAM is comprised of 22 evaluation items within the 6 original categories. The SMOG is a readability assessment tool that uses a formula to calculate grade levels by the number of sentences, total number of words in the sentences, and the number of polysyllabic words
  Arms: Samoan Original Assessment Tools
Behavioral: CDC Colorectal cancer screening for life brochure: SAM + CAM Cloze Procedure — Suitability and Comprehensibility Assessment of Materials (SAM + CAM). The SAM + CAM is comprised of 22 evaluation items within the 6 original categories. The SMOG is a readability assessment tool that uses a formula to calculate grade levels by the number of sentences, total number of words in the sentences, and the number of polysyllabic words
  Arms: Samoan Original Assessment Tools
Behavioral: Colocare Instruction Sheet: SAM + CAM - Superior rating Cloze Procedure — Suitability and Comprehensibility Assessment of Materials (SAM + CAM). The SAM + CAM is comprised of 22 evaluation items within the 6 original categories. The SMOG is a readability assessment tool that uses a formula to calculate grade levels by the number of sentences, total number of words in the sentences, and the number of polysyllabic words
  Arms: Samoan Modified Assessment Tools
Behavioral: CDC Colorectal Cancer Screening for Life Brochure: SAM + CAM - Superior rating Cloze Procedure — Suitability and Comprehensibility Assessment of Materials (SAM + CAM). The SAM + CAM is comprised of 22 evaluation items within the 6 original categories. The SMOG is a readability assessment tool that uses a formula to calculate grade levels by the number of sentences, total number of words in the sentences, and the number of polysyllabic words
  Arms: Samoan Modified Assessment Tools

SUMMARY:
This study, led by the American Samoa Community Cancer Coalition's INdigenous Samoan Partnership to Initiate Research Excellence (INSPIRE) and the UH Cancer Center's project team including Dr. Cassel, will utilize a community-based and culturally relevant process to assess the uptake of fecal occult blood testing (FOBT) using tailored colorectal cancer patient education materials for those with inadequate health literacy. Our primary outcomes include: 1) process to develop "suitable" and "comprehensible" health promotion materials for populations in English and Samoan with various health literacy levels, 2) commitment to use the FOBT Colocare home kit, and 3) use of a FOBT Colocare home kit.

DETAILED DESCRIPTION:
Utilizing the Behavioral Model of Health Services Use as a conceptual framework and the evidence-based program "Against Colorectal Cancer in Our Neighborhoods" (ACCION) for the Latino population in Texas as a guide, the proposed study will conduct a randomized controlled trial of Indigenous Samoan participants (N=312), age≥ 50 recruited using Respondent-Driven Sampling (RDS). This design will compare use of non-tailored instruction for completing ColoCare FOBT home-kits (N=156) versus the experimental condition, using a ColoCare FOBT home-kit with instructions tailored to low health literacy and to enhance CRC-Knowledge Attitudes and Behavior (KAB) - (N=156). Our goal is to test the influence of tailored materials on timely completion of CRC screening using the ColoCARE FOBT.

ELIGIBILITY:
Inclusion Criteria:

1. Resident of America Samoa
2. Over age 50
3. Have not been diagnosed or treated for colon cancer
4. Is not high risk for CRC by having family history or diagnosed with irritable bowel syndrome
5. Can read and speak English and Samoan (can provide written informed consent)
6. Have a home address and working phone
7. Is willing to provide information on their health behaviors

Exclusion Criteria:

* persons who indicate they speak or read and write Samoan or English less than well

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Tofaeono, M.D., Principal Investigator — American Samoa Community Cancer Coalition
Locations (2):
- American Samoa (2):
  - American Samoa Community Cancer Coalition, Pago Pago
  - American Samoa Power Authority Abe Malae Operations Center, Tafuna

IPD SHARING:
Plan to Share IPD: Yes
Study data will be administered in accordance with UHCC policies. Data will be accessible only to study staff. Study staff includes Principal Investigators, Project Director, and Researchers.
  Upon completion community members and partners will have access to aggregated data. After data analysis is completed, study materials will be kept in the PI's locked office and destroyed after five years. The data and associated documentation will be available to the study team only under a data-sharing agreement that provides for: a commitment to using the data only for research purposes and not to identify any individual participant, a commitment to securing the data using appropriate computer technology, and a commitment to destroying the data after analyses are completed. The products/resources that result of this study will be disseminated via publications, presentations at national conferences, presentations, and reports to study stakeholders.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: September 2020
Access Criteria: Data will be accessible only to the study staff to ensure confidentiality. Study staff includes Principal Investigators, Project Director, and Researchers.
  Upon completion community members and partners such as the Department of Health, Lyndon B. Johnson Tropical Medical Center, and the Cancer Council of the Pacific Islands will have access to aggregated data

REFERENCES:
- [Background] American Samoa Department of Health (2013). Behavioral Risk Factor Surveillance Survey. Results and Data Report. Fagaalu, American Samoa
- [Background] Efird J. Blocked randomization with randomly selected block sizes. Int J Environ Res Public Health. 2011 Jan;8(1):15-20. doi: 10.3390/ijerph8010015. Epub 2010 Dec 23. PMID 21318011
- [Background] Walter SD, Eliasziw M, Donner A. Sample size and optimal designs for reliability studies. Stat Med. 1998 Jan 15;17(1):101-10. doi: 10.1002/(sici)1097-0258(19980115)17:13.0.co;2-e. PMID 9463853
- [Background] Johnston LG. Introduction to respondent-driven sampling. Technical report. 2008 http://bit.ly/OHgGX5

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | English Original Assessment Tools | Samoan Original Assessment Tools | English Modified Assessment Tools | Samoan Modified Assessment Tools
Started | 58 | 90 | 40 | 76
Completed | 58 | 90 | 40 | 76
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | English Original Assessment Tools | Samoan Original Assessment Tools | English Modified Assessment Tools | Samoan Modified Assessment Tools | Total
Number analyzed (Participants) | 58 | 90 | 40 | 76 | 264
Age, Categorical [Count of Participants; unit: Participants] — Population: Unknown birth year for 11 participants
  Participants
    number analyzed (Participants) | 56 | 87 | 37 | 73 | 253
    <=18 years | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 52 | 80 | 32 | 66 | 230
    >=65 years | 4 | 7 | 5 | 7 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 67 | 30 | 16 | 157
  Male | 14 | 23 | 10 | 60 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 58 | 90 | 40 | 76 | 264
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 57 | 90 | 38 | 76 | 261
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  American Samoa | 58 | 90 | 40 | 76 | 264

OUTCOME MEASURES:

1. Primary Outcome: Use of FOBT ColoCARE Home Kit
Description: Number of participants reporting results for the FOBT ColoCARE Home kit
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | English Original Assessment Tools | Samoan Original Assessment Tools | English Modified Assessment Tools | Samoan Modified Assessment Tools
Number analyzed (Participants) | 58 | 90 | 40 | 73
participants | 14 | 2 | 14 | 0

2. Primary Outcome: Increase Uptake of FOBT ColoCARE Home Kit
Description: Change in CRC-Knowledge Attitudes and Behavior (KAB) among subjects who viewed the tailored ColoCARE video. This measure is a 7 question assessment given before and after participants viewed the ColoCARE video. Participants were scored based on their pre and post assessment responses.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | English Original Assessment Tools | Samoan Original Assessment Tools | English Modified Assessment Tools | Samoan Modified Assessment Tools
Number analyzed (Participants) | 58 | 90 | 40 | 73
Participants
  Positive Change | 48 | 84 | 23 | 67
  Negative Change | 10 | 6 | 17 | 6

3. Primary Outcome: Modified Patient Education Materials
Description: Use a combination of inadequate health literacy recommendations, suitable, and comprehensible assessment methods to develop modified culturally appropriate patient education materials for Colorectal Cancer (CRC). Each of the 22 items within the 6 identified categories are given a score of 0 - 2 based upon certain criteria. Total scores are calculated into percentages and 100% to 70% is "adequate", "69% to 40%" is "marginal, while 39% - 0% is "inadequate".
Time Frame: 1 Month
Measure: Count of Participants; unit: Participants
Arm/Group | English Original Assessment Tools | Samoan Original Assessment Tools | English Modified Assessment Tools | Samoan Modified Assessment Tools
Number analyzed (Participants) | 58 | 90 | 40 | 73
Participants
  Adequate STOFHLA Score | 41 | 18 | 27 | 10
  Marginal STOFHLA Score | 13 | 25 | 9 | 26
  Inadequate STOFHLA Score | 4 | 47 | 4 | 37

ADVERSE EVENTS:
Time Frame: The incidence and severity of adverse events occurring during the study intervention will be reported. Subjects participated in the study for 3 weeks maximum, with the total study reporting period lasting from 9/2020 until 1/2021.
Description: This is a minimal risk study, and we do not anticipate serious adverse events or mortality.
Arm/Group | English Original Assessment Tools | Samoan Original Assessment Tools | English Modified Assessment Tools | Samoan Modified Assessment Tools
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/90 | 0/40 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/90 | 0/40 | 0/76
Other Adverse Events (participants affected / at risk) | 0/58 | 0/90 | 0/40 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/71/NCT04500171/Prot_ICF_000.pdf